CLINICAL TRIAL: NCT00668538
Title: Uptake of the Antifungal Miconazole and Effect on Estrogen Metabolizing Enzymes in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Professor, M.D. Kim Brosen, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AKF-373; EudraCT 2008-000796-17
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Miconazole; CYP1A2; CYP3A4; Women; Healthy Subjects
MeSH Terms: interventions — Miconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Brentan (miconazole) — Vaginal suppository 1200 mg at day 6
  Other Names: miconazole

SUMMARY:
The purpose of this study, is to study the uptake of the pharmaceutical antifungal miconazole when used as a vaginal suppository in young women. The investigators want to know if the uptake is big enough to cause a biological effect (effect on CYP1A2 and CYP3A4 activity).

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Age 18-45 years
* Healthy
* Signed consent
* Written authority to the GCP-unit

Exclusion Criteria:

* Pregnancy
* Breast-feeding
* Hypersensitivity to miconazole
* Hypersensitivity to sodium ethyl parahydroxybenzoic acid(E219)
* Hypersensitivity to sodium propyl parahydroxybenzoic acid (E217)
* Using contraceptives with hormones
* Daily consumption of alcohol
* Daily use of medicine
* Participated in a clinical trial within the last 3 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
CYP1A2 and CYP3A4 activity measured as metabolite ratios of caffeine and quinidine, respectively | urine and blood collected day 4 and 8

SECONDARY OUTCOMES:
Detection of miconazole or metabolites in blood and urine | Blood and urine collected day 8

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Public Health, Clinical Pharmacology, University of Southern Denmark, Odense, Denmark

REFERENCES:
- [Derived] Kjaerstad MB, Nielsen F, Nohr-Jensen L, Zwisler S, Brosen K, Andersen HR. Systemic uptake of miconazole during vaginal suppository use and effect on CYP1A2 and CYP3A4 associated enzyme activities in women. Eur J Clin Pharmacol. 2010 Dec;66(12):1189-97. doi: 10.1007/s00228-010-0906-2. Epub 2010 Oct 6. PMID 20924570